CLINICAL TRIAL: NCT06881732
Title: Experimental Malaria Infection of Healthy Malaria-Naive Adults by Mosquito Bite With the Genetically Modified Plasmodium Falciparum NF54/iGP3 GAP
Acronym: iGP3-SWITCH
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other); Swiss Tropical & Public Health Institute (Other); QIMR Berghofer Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UoM/DCT/2024-02
Record Dates: First submitted 2025-02-27; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Malaria Falciparum; Malaria Infection; Malaria Transmission
Keywords: SWITCH; NF54/iGP3; Plasmodium falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: All participants enrolled into the study will be infected with the malaria parasite.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Plasmodium falciparum NF54/iGP3 (Experimental): Infection by direct feeding of Anopheles stephensi mosquitoes infected with Plasmodium falciparum NF54/iGP3
  Interventions: Biological: NF54/iGP3

INTERVENTIONS:
Biological: NF54/iGP3 — Mosquito-generated sporozoites of the genetically modified, inducible gametocyte-producing parasite line NF54/iGP3, created via CRISPR/Cas9 genetic engineering of the parental wildtype strain Plasmodium falciparum (Pf) NF54 to contain a trimethoprim (TMP)-inducible copy of the Pf gdv1 gene in the dispensable Pf cg6 locus.

SUMMARY:
The goal of this clinical trial is to learn if the genetically-modified malaria parasite NF54/iGP3 will safely infect humans with malaria. The investigators will also determine how the parasite grows in humans, and the effect of anti-malarial drugs.

Researchers will use a controlled human malaria infection (CHMI) model to infect participants with malaria to observe the development of the disease, collect malaria-infected blood, and then treat the participants to cure the malaria infection.

The collected malaria-infected blood will be used to create a frozen stock of malaria parasites for use in future research.

DETAILED DESCRIPTION:
Malaria is caused by the Plasmodium parasite and is spread through the bite of mosquitos. During the blood stage of a malaria infection, the parasite can be found in four different forms. Most antimalarial drugs effectively kill the parasites, however, they do not kill one form of the parasite known as gametocytes. Gametocytes are important in the spread of malaria as they are the only form which can be passed from human back to a mosquito.

Currently, primaquine (an antimalarial drug) is the only medicine which kills gametocytes. However, this cannot be given to everyone. Individuals with certain genetic and metabolic disorders, including glucose-6-phosphate dehydrogenase (G6PD) deficiency, face severe health risks if they take Primaquine. Testing for G6PD deficiency is expensive and not available worldwide, which further reduces the number of individuals who can safely take this medication. Therefore, researchers need to develop new antimalarial drugs which kill gametocytes that are safe for all people.

Developing an improved controlled human malaria infection (CHMI) model which produces more gametocytes is a crucial step in advancing antimalarial research, especially targeting the transmission stage. To achieve this, the investigators have created a laboratory made genetically modified (change in DNA), malaria parasite known as Plasmodium falciparum NF54/iGP3, which makes an increased number of gametocytes in comparison with naturally occurring malaria parasites.

The purpose of this study is to develop a CHMI with NF54/iGP3 genetically altered parasites to assess the safety of infecting humans with this malaria parasite as well as determine the growth of the malaria parasites in humans and the effect of anti-malarial drugs. Samples from this study will be used to create a master cell bank of the NF54/iGP3 parasite, so that future research can be carried out using a malaria blood-stage infection model that will produce a greater proportion of gametocytes during infection.

The importance of this research is crucial for the future development and testing of new treatments and vaccines against malarial gametocytes. The development of new antimalarial drugs against malarial gametocytes will over time prevent malaria being transmitted from humans to mosquitos ultimately eliminating the continual spread of malaria.

ELIGIBILITY:
INCLUSION CRITERIA:

* Able and willing to complete the informed consent process
* Available for the entire planned study duration
* Male or Female
* Aged 18 to 55 years
* Willing to have blood samples collected, stored indefinitely and used for research purposes
* Willing to defer blood donations for at least six months after the EoS visit (D180)
* Agreement to adhere to specific Lifestyle Considerations throughout study duration

Clinical Criteria:

* Total body weight ≥ 50 kg, and a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive)
* In good general physical and mental health as evaluated through a comprehensive clinical assessment
* Vital signs at screening and pre-inoculation within normal clinical range
* Electrocardiograph (ECG) without significant abnormalities, including: QTcF ≤450 ms for males, QTcF ≤470 ms for females, PR interval ≤210 ms

Laboratory Criteria:

* O negative blood type
* Haemoglobin, white cell count and platelet levels within normal laboratory ranges
* Ferritin, creatinine and alanine aminotransferase (ALT) within normal laboratory ranges
* No clinically significant abnormality in coagulation or clotting
* Normal G6PD enzyme activity levels as defined by the parameters of the specific quantitative G6PD test performed at screening
* Negative for blood borne viruses, including Human Immunodeficiency Virus (HIV), Hepatitis B virus (HBV), Hepatitis C virus (HCV), Human T-lymphotropic virus type 1 (HTLV); and other blood borne pathogens including West Nile Virus (WNV), Babesia species, Treponema pallidum, and Trypanosoma cruzi

Criteria specific to female participants:

* Post-menopausal for at least 1 one year, post-hysterectomy, or bilateral oophorectomy with a correlating follicle stimulating hormone (FSH) level.

OR

* Females of childbearing age have a negative beta-human chorionic gonadotrophin (b-HCG) pregnancy test (urine or serum) on day of enrolment and prior to CHMI inoculation and agreement to use effective birth control through the duration of the study.

EXCLUSION CRITERIA:

* Participant lives alone and is unable provide contact details of a support person who is aware of the individual's participation in the study and is available to provide assistance if required
* Participation in any investigational product study within the 12 weeks preceding inoculation
* Positive urine drug test at screening or on the day of malaria inoculation unless there is an explanation acceptable to the Investigator (e.g. the volunteer has stated in advance that they consumed a prescription or over-the-counter product which contained the detected drug) and/or the volunteer has a negative urine drug screen on retest by the pathology laboratory
* Positive alcohol breath test at screening or on the day of malaria inoculation

Malaria History:

* Any previous history of malaria infection, including participation in a malaria research study
* Receipt of a malaria vaccination at any time, including as part of a research study
* Travelled to or lived (more than two weeks) in a malaria-endemic region during the past 12 months or planned travel to a malaria-endemic region over the course of the study
* Lived for more than one year in a malaria-endemic region in the past 10 years
* Lived in a malaria-endemic region for more than 10 years inclusive

Clinical History:

* Anyone who is pregnant, breastfeeding or planning pregnancy during the study period
* History of severe allergic reaction, including angioedema or anaphylaxis
* Receipt of any live attenuated vaccines within 21 days prior to enrolment
* Has ever received a blood transfusion
* Use of blood products or immunoglobulins within the previous 6 months
* Without good peripheral venous access
* Clinical history of: Sickle cell disease, sickle cell trait or other haemoglobinopathies; Splenectomy or fuctional asplenia; Skeeter syndrome or anaphylactic response to mosquito bites
* Known intolerance, hypersensitivity or other contraindication to artemether or other artemisinin derivatives, lumefantrine, atovaquone, proguanil, primaquine, or artesunate or any of its excipients
* Use or planned use of any drug, including antibiotics, with antimalarial activity four weeks prior to inoculation
* Use of any of the following drugs: Anticoagulants (within 14 days of enrolment); Systemic corticosteroids (within 3 months of enrolment); Any prescription or non-prescription drugs, and or supplements that in the opinion of the investigator would jeopardise the safety of the volunteer
* Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer, including but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, autoimmune disease, infectious diseases, psychiatric disorders, heart disease, or cancer

Clinical Risk:

* Evidence at screening of increased cardiovascular disease risk (defined as >10%, 5-year risk for those greater than 35 years of age), as determined by the Australian Absolute Cardiovascular Disease Risk Calculator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To assess the infectivity, safety and tolerability of mosquito bite sporozoite challenge with NF54/iGP3 in healthy malaria-naïve participants by counting solicited and unsolicited adverse events. | From Inoculation (Day 1) until End of Study (Day 180)
  Count the occurrence and assess the severity of local and systemic, solicited and unsolicited adverse events using CTCAE v5.0, following administration of NF54/iGP3 by mosquito bite.

SECONDARY OUTCOMES:
To characterise the parasite growth profile of all blood stage parasites in participants following infection with NF54/iGP3 using qPCR (parasites/mL). | From Inoculation (Day 1) until conditions for treatment are met (truncated at Day 22)
  Measure the change in parasite count (parasites/mL) of blood-stage NF54/iGP3 parasites via qPCR, following inoculation until the administration of antimalarial treatment.
To characterise the post-treatment clearance profile of all blood stage parasites in participants following infection with NF54/iGP3 using qPCR (parasites/mL). | From administration of antimalarial treatment until End of Study (Day 180)
  Measure the change in parasite count (parasites/mL) of blood-stage NF54/iGP3 parasites via qPCR, following administration of registered schizonticidal and gametocidal antimalarial treatments.
Measure the parasite count (parasites/mL) using qPCR in the participant's blood at the time of large volume blood withdrawal. | From Inoculation (Day 1) until parasitemia conditions are met, truncated at Day 22
  Measure the parasite count (parasites/mL) via qPCR in collected blood samples from study participants infected with NF54/iGP3, to determine the level of parasitemia.

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Principal Investigator — University of Melbourne
Locations (1):
- Doherty Clinical Trials, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided